CLINICAL TRIAL: NCT07091500
Title: Effect of GLP-1 Receptor Agonist Therapy With and Without Exercise Training on Muscle Mass and Physical Function in People With Obesity
Brief Title: Glucagon-like Peptide 1 (GLP-1) Receptor Agonist Therapy and Exercise Training in People With Obesity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 202505162
Record Dates: First submitted 2025-07-10; First posted 2025-07-29 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Obesity; Skeletal Muscle
MeSH Terms: conditions — Obesity | interventions — Exercise; semaglutide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GLP-1 RA (Active Comparator): Participants in this group will receive semaglutide therapy along with diet behavior counseling for 52 weeks
  Interventions: Drug: Semaglutide
- GLP-1 RA + Exercise (Experimental): Participants in this group will receive semaglutide therapy along with diet behavior counseling and exercise training for 52 weeks.
  Interventions: Behavioral: Exercise training; Drug: Semaglutide

INTERVENTIONS:
Behavioral: Exercise training — Participants will perform supervised exercise training sessions 3 days per week and unsupervised at-home sessions 2-3 days per week.
  Arms: GLP-1 RA + Exercise
Drug: Semaglutide — semaglutide 2.4 mg subcutaneous per week or max tolerated dose and diet behavior counseling

SUMMARY:
The use of glucagon-like peptide receptor agonists (GLP-1 RAs) may have clinically important effects on skeletal muscle mass (SMM), and physical function. The effects of exercise training in conjunction with GLP-1 RA therapy on these outcomes has not been studied. Additionally, most people treated with GLP-1-based weight loss medications stop taking these medications within 1 year of initiating treatment. This is an important clinical concern because weight regain can occur after weight loss pharmacotherapy is stopped and the impact of stopping GLP-1 RA therapy on physical and metabolic function has not been studied.

In this study, the investigators will conduct a 2-year randomized clinical trial to evaluate body composition, muscle physical and metabolic function, and muscle strength in response to GLP-1 RA therapy, with or without exercise training, and subsequent treatment cessation on muscle-related outcomes.

ELIGIBILITY:
Inclusion Criteria:

* i) obesity (Body Mass Index ≥ 30 kg/m2)
* ii) decreased physical function (Modified Physical Performance Test score 17 to 31)
* iii) approval of their primary physician to participate in this study.

Exclusion Criteria:

* i) unstable weight (>4% change during the last 2 months before entering the study)
* ii) ≥150 min per week of structured exercise (e.g., jogging, activities that cause heavy breathing and sweating)
* iii) diabetes
* iv) significant cardiopulmonary disease (heart failure, angina, uncontrolled hypertension, chronic obstructive pulmonary disease) or other organ dysfunction (e.g., renal insufficiency [eGFR <30 mL/min/1.73 m2])
* v) therapy with a GLP-1 or other weight loss medications
* vi) clinically significant gastric emptying abnormality or chronically take drugs that directly affect gastrointestinal motility
* vii) history of chronic or acute pancreatitis
* viii) thyroid-stimulating hormone (TSH) >1.5X the upper limit of normal (patients receiving treatment for hypothyroidism may be included provided their thyroid hormone replacement dose has been stable for at least 3 months)
* ix) history of significantly active or unstable Major Depressive Disorder or other severe psychiatric disorder (e.g. schizophrenia, bipolar disorder, or other serious mood or anxiety disorder) within the last 2 months that would interfere with study participation
* x) acute or chronic hepatitis, or other liver disease other than Metabolic dysfunction-Associated Steatotic Liver Disease (MASLD)
* xi) family or personal history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome type 2
* xii) history of active or untreated malignancy or are in remission from a clinically significant malignancy (other than basal- or squamous cell skin cancer, in situ carcinomas of the cervix, or in situ prostate cancer) for less than 5 years
* xiii) tobacco use, excessive alcohol intake (≥3 drinks/day for men and ≥2 drinks/day for women) or active substance abuse with illegal drugs by self-report, or regular marijuana use within 3 months of enrollment and unwilling to abstain from marijuana during the trial
* xiv) Use of medications that are known to affect the study outcome measures or increase the risk of study procedures and that cannot be temporarily discontinued for this study
* xv) have had bariatric surgery or plan to have endoscopic or bariatric surgery therapy for obesity
* xvi) anemia (Hgb <10 g/dL)
* xvii) Conditions that render subject unable to complete all testing procedures (e.g., severe ambulatory impairments, limb amputations, or metal implants that interfere with imaging procedures; coagulation disorders)
* xii) history of seizure disorder
* xix) Female who is pregnant, breast-feeding or intends to become pregnant
* xx) allergy or hypersensitivity to GLP-1 RA medications
* xxi) unable to grant voluntary informed consent
* xxii) unable or unwilling to follow the study protocol or who, for any reason, the research team considers the participant is not an appropriate candidate for the study

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-11 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Physical function | Baseline, after 52 weeks of intervention, and 52 weeks after stopping the intervention
  Score on the Modified Physical Performance Test
Body composition | Baseline, after 52 weeks of intervention, and 52 weeks after stopping the intervention
  DEXA scan

SECONDARY OUTCOMES:
Muscle mass | Baseline, after 52 weeks of intervention, and 52 weeks after stopping the intervention
  Whole-body muscle mass will assessed by using the D3-creatine dilution method
Muscle volume | Baseline, after 52 weeks of intervention, and 52 weeks after stopping the intervention
  Magnetic resonance scans
Insulin sensitivity | Baseline, after 52 weeks of intervention, and 52 weeks after stopping the intervention
  Whole-body insulin sensitivity during a hyperinsulinemic-euglycemic clamp
Muscular Strength for the Chest Press exercise | Baseline, after 52 weeks of intervention, and 52 weeks after stopping the intervention
  Upper body muscle strength will be assessed as a ten repetition maximal strength for the chest press exercise on a Hoist multi-station weight machine
Muscular Strength for the Seated Row exercise | Baseline, after 52 weeks of intervention, and 52 weeks after stopping the intervention
  Upper body muscle strength will be assessed as a ten repetition maximal strength for the seated row exercise
Muscular Strength for the Leg Press exercise | Baseline, after 52 weeks of intervention, and 52 weeks after stopping the intervention
  Lower body muscle strength will be assessed as a ten repetition maximal strength for the leg press exercise
Muscular Strength for the Leg Flexion exercise | Baseline, after 52 weeks of intervention, and 52 weeks after stopping the intervention
  Lower body muscle strength will be assessed as a ten repetition maximal strength for the leg flexion exercise

CONTACTS AND LOCATIONS:
Overall Officials: Joseph W Beals, PhD, Study Director — Washington University School of Medicine; Samuel Klein, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States